CLINICAL TRIAL: NCT03475316
Title: Social Dancing Intervention for Older Adults at High Risk of Alzheimer's Disease and Other Dementias: A Pilot Study.
Brief Title: Movement Intervention for Memory Enhancement
Acronym: MIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Joe Verghese, Professor of Neurology & Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-8942; 1R21AG057586-01A1 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-03-23 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease; Dementia; Cognitive Decline; Cognitive Impairment; Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Dancing (Experimental): The program includes Fox-trot, Waltz, and Latin dances.
  Interventions: Behavioral: Social Dancing
- Treadmill Walking (Active Comparator): The treadmill walking training protocol is based on the recommendations of the American College of Sports Medicine (ACSM) and American Heart Association (AHA) for older adults.
  Interventions: Behavioral: Treadmill Walking

INTERVENTIONS:
Behavioral: Social Dancing — 90-min dance sessions twice weekly for 6-months. The session includes warm-up, dance and cool down.
  Arms: Social Dancing
Behavioral: Treadmill Walking — Each session starts with 5-10 minutes of warm-up walking at comfortable speed. Speed is gradually increased to the level at which participants felt it is 'somewhat hard' for two 35 minute sessions with breaks in between followed by 5-10 minute cool down period (total 90 min to match dance group).
  Arms: Treadmill Walking

SUMMARY:
Dancing is a complex sensorimotor rhythmic activity that integrates cognitive, physical, and social components and is applicable to seniors with various fitness levels. Despite its popularity, there is a paucity of studies that have systematically examined the role of dancing in preventing or delaying cognitive decline in older adults at high risk for Alzheimer's disease and related dementias. This preliminary randomized clinical trial will help provide the evidence base to develop a definitive full-scale trial to support or refute prescription of social dancing to prevent further cognitive decline in older adults at high risk of Alzheimer's disease and related dementia.

DETAILED DESCRIPTION:
Social dancing is a complex sensorimotor rhythmic activity integrating physical, cognitive and social elements with the potential to ameliorate a wide range of physical and cognitive impairments in older individuals at risk of Alzheimer's disease (AD) and related dementias. The few extant studies report that dancing stimulates multiple cognitive processes, including attention, processing speed, and executive function, but these discoveries were made in small samples, lacking control conditions, and did not investigate the underlying biological mechanisms.

Executive function (EF) is an umbrella term for the management of cognitive processes, including working memory, reasoning, task flexibility, and problem solving that are central to planning, goal-directed action, and coordination of daily activities. Impairment of EF and related processes such as processing speed and attention is seen in normal aging as well as early in dementia, and is associated with difficulty in performing daily activities and increased risk of adverse events such as falls. Encouragingly, aerobic exercise is reported to enhance cognition, especially EF. Cognitively impaired seniors fall more, and have higher prevalence and severity of balance and gait problems than cognitively intact fallers. Given social dancing's multimodal cognitive and physical benefits; it may help maintain mobility and reduce falls in individuals at risk for dementia. In support, the investigators reported that older social dancers had better balance and gait than non-dancers.

The investigators propose a 6-month pilot single blind, randomized clinical trial (RCT) comparing social dancing (ballroom dancing) versus active control (walking) in 32 older adults at high risk of dementia. The overall hypothesis is that social dancing in cognitively vulnerable seniors will induce neuroplasticity that will enhance cognitive processes and improving everyday behaviors. The objective for this pilot trial is to obtain preliminary data on intervention effects (trajectory and asymptote) on EF to design a full-scale RCT.

Social dancing appeals to older adults, has intrinsic value, is enjoyable, and has high potential for sustainability. This trial is novel and high risk, but will provide the evidence base to develop a definitive full-scale RCT to support or refute prescription of social dancing to prevent cognitive decline in older adults at high risk of AD and related dementias.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 and older
* A score of ≤ 6 on the Memory Impairment Screen or ≥ 1 on the AD-8
* Plan to be in area for next year or more
* English speaking
* Willing to complete an Functional Magnetic Resonance Imaging (MRI)

Exclusion Criteria:

* Presence of dementia based on previous physician diagnosis of dementia or dementia diagnosed by the study clinician at initial visit.
* Serious chronic or acute illness such as cancer (late stage, metastatic, or on active treatment), chronic pulmonary disease on ventilator or continuous oxygen therapy or active liver disease.
* Mobility limitations solely due to musculoskeletal or cardiovascular conditions that prevent participation in the intervention programs.
* Any medical condition or chronic medication use (e.g., neuroleptics) in the judgment of the screening clinician that will compromise safety or affect cognitive functioning.
* Terminal illness with life expectancy less than 12 months.
* Presence of progressive, degenerative neurologic disease (e.g., Parkinson's disease or Amyotrophic lateral sclerosis).
* Severe auditory or visual loss.
* Active psychoses or psychiatric symptoms (such as agitation) noted during the clinic visit that will prevent completion of study protocols.
* Either participation in competitive dancing or recreational dancing at a frequency >1/month in the past six months.
* Participation in other interventional study that overlaps with intervention period of this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MBBS, Principal Investigator — Albert Einstein College of Medicine; Helena Blumen, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumen HM, Ayers E, Wang C, Ambrose AF, Verghese J. A social dancing pilot intervention for older adults at high risk for Alzheimer's disease and related dementias. Neurodegener Dis Manag. 2020 Aug;10(4):183-194. doi: 10.2217/nmt-2020-0002. Epub 2020 Aug 3. PMID 32741240

RESULTS

PARTICIPANT FLOW:
Period: 6 Month Intervention
Arm/Group | Social Dancing | Treadmill Walking
Started | 13 | 12
Completed | 8 | 8
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study stopped due to COVID pandemic | 1 | 3
Period: 9 Months
Arm/Group | Social Dancing | Treadmill Walking
Started | 8 | 8
Completed | 5 | 4
Not Completed | 3 | 4
Not completed — Study stopped due to COVID pandemic | 3 | 4

BASELINE CHARACTERISTICS:
Population: Includes all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Dancing | Treadmill Walking | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (5.82) | 75.43 (5.84) | 76.45 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 7 | 5 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Years of education [Mean (Standard Deviation); unit: years] | 16.62 (4.61) | 14.67 (4.23) | 15.68 (4.51)

OUTCOME MEASURES:

1. Primary Outcome: Executive Function (EF).
Description: Improvement in EF will be measured through a composite score from 3 tests. (1) The Digit Symbol Substitution test is a measure of attention and speed of processing. Scoring is based on the total number of correct responses generated over 90 seconds. Higher values reflect better outcome. (2) Flanker Test is a measure of speed of processing, attention and inhibitory control. Scoring is based on accuracy and reaction time. Lower values reflect better outcome. (3) Walking While Talking (repeating alternating letters of the alphabet) gait speed (centimeters/second) will be measured using a electronic walkway system. Higher values reflect better outcome. The scores on the 3 tests are standardized and summed to obtain a single z-score. The Z-score indicates the number of standard deviations away from the mean of the study population and a value of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean.
Time Frame: Baseline, 6 months
Population: Includes all participants who were randomized except 3 participants in the Treadmill walking group who were missing 1 or more of the 3 composite score tests.
Measure: Mean (Standard Error); unit: z score
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 13 | 9
z score | 1.16 (0.42) | 0.99 (0.39)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Linear mixed effects model were used to compare changes in the composite score pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-1.14 to 1.49], Standard Error of Mean 0.57 — The estimate parameter is the difference in change at post intervention from pre between dance and treadmill group

2. Secondary Outcome: Neuroplasticity.
Description: Functional Magnetic Resonance Imaging will be used to investigate neuroplasticity under three conditions: 'imagined Walking While Talking' task, Digit Symbol Substitution test and Flanker interference tests. Functional activation/deactivation patterns recorded by Functional Magnetic Resonance Imaging in response to the three tests will be examined within each participant before and after the intervention. The values measured as factor scores reflect change in functional activation/deactivation covariance patterns from pre to post intervention as a function intervention (social dancing vs. treadmill walking). Larger absolute values reflect more change in functional activation/deactivation covariance patterns from pre to post intervention on each of the three tasks. There is no set minimum and maximum values of the scale.
Time Frame: Baseline, 6 months
Population: Includes all participants who completed the baseline MRI session and was randomized, except 3 participants in the Social Dancing group and 2 participants in the Treadmill Walking group with incomplete tasks/session or corrupted data files.
Measure: Mean (Standard Error); unit: units on a scale (factor scores)
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 9 | 6
units on a scale (factor scores)
  functional activation/deactivation covariance patterns during Digit Symbol Substitution test | -9.68 (170.38) | -273.47 (492.47)
  functional activation/deactivation covariance patterns during Flanker Interference test | 6.82 (30.98) | -17.44 (53.73)
  functional activation/deactivation covariance patterns during imagined Walking While Talking | 81.30 (63.16) | 21.94 (106.65)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Estimates with standard errors (SE) are from linear mixed effect models used to examine the difference in change in functional activation/deactivation covariance patterns during the Digit Symbol Substitution test at post intervention from pre intervention between the social dancing and treadmill walking group; Test type: Superiority; Mean Difference (Net) = 166.16, 95% CI 2-sided [-231.12 to 563.44], Standard Error of Mean -202.70 — The estimate parameter reflects change in functional activation/deactivation pattern from pre to post intervention as a function intervention (social dancing vs. treadmill walking)
Statistical Analysis 2: Comparison: Social Dancing vs Treadmill Walking; Estimates with standard errors (SE) and p-values are from linear mixed effect models used to examine the difference in change in functional activation/deactivation covariance patterns during the Flanker interference test at post intervention from pre intervention between the social dancing and treadmill walking group; Test type: Superiority; Mean Difference (Net) = 24.60, 95% CI 2-sided [-31.20 to 80.40], Standard Error of Mean 28.47 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Social Dancing vs Treadmill Walking; Estimates with standard errors (SE) are from linear mixed effect models used to examine the difference in functional activation/deactivation covariance patterns during the Imagery of Walking-While Talking task at post intervention from pre intervention between the social dancing and treadmill walking group; Test type: Superiority; Mean Difference (Net) = 58.22, 95% CI 2-sided [-42.14 to 158.58], Standard Error of Mean 51.20 — [estimate comment as in outcome 2, analysis 1]

3. Other Pre Specified Outcome: Lifestyle Changes.
Description: Lifestyle changes will be measured at baseline and post-intervention through the Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire. CHAMPS scale measures weekly frequency/week of moderate-intensity exercise-related activities. Scores range from 0 to 133 with higher score indicating more exercise
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 13 | 12
score on a scale | 0.41 (1.09) | -0.36 (2.47)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Linear mixed effects model were used to compare changes in the CHAMPS scores pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-5.10 to 6.64], Standard Error of Mean 2.70 — The Estimation Parameter is the difference in change at post from pre between dance and treadmill group

4. Other Pre Specified Outcome: Gait.
Description: Changes in gait speed will be measured at baseline and post-intervention through a quantitative gait mat. Gait is measured in centimeters per second and higher values indicate faster walking speed.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: centimeters per second
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 13 | 12
centimeters per second | 11.39 (7.26) | 4.11 (4.56)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Linear mixed effects model were used to compare changes in gait speed pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 7.27, 95% CI 2-sided [-11.60 to 26.14], Standard Error of Mean 8.57 — The estimate parameter is the difference in change at post intervention from pre between dance and treadmill group

5. Other Pre Specified Outcome: Balance
Description: Changes in balance will be measures at baseline and post-intervention using the Unipedal stance (measured in seconds). Higher time indicates better balance.
Time Frame: Baseline, 6 months
Population: Includes all randomized participants, but excludes 8 participants in the experimental group who were unable to do the assessment.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 8 | 12
seconds | 2.03 (4.72) | 1.46 (3.55)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Linear mixed effects model were used to compare changes in unipedal stance time pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-13.40 to 14.55], Standard Error of Mean 5.91 — The estimate parameter is the difference in change at post intervention from pre between dance and treadmill group

6. Other Pre Specified Outcome: Modified Katz Disability Scale.
Description: Changes in function assessed by 4 key activities of daily living tasks-bathing, dressing, walking, and transferring. Scores range from 0 to 8 with higher scores indicating worse outcome.
Time Frame: Baseline, 6 months
Population: This measure was not completed; therefore, no outcome data is included.
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: The Geriatric Depression Scale (GDS).
Description: Changes in depressive symptoms assessed using the 30 item GDS, scores range from 0 (not depressed) to 30 (depressed).
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Social Dancing | Treadmill Walking
Number analyzed (Participants) | 13 | 12
score on a scale | 1.41 (0.55) | 0.33 (0.96)
Statistical Analysis 1: Comparison: Social Dancing vs Treadmill Walking; Linear mixed effects model were used to compare changes in the geriatric depression scale pre and post intervention; Test type: Superiority; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [-1.30 to 3.46], Standard Error of Mean 1.11 — The estimate parameter is the difference in change at post intervention from pre between dance and treadmill group

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Social Dancing | Treadmill Walking
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Dancing (N=13) | Treadmill Walking (N=12)
Falls (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
High blood pressure (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03475316/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03475316/ICF_001.pdf